CLINICAL TRIAL: NCT01602458
Title: The Use of Pressure and Silicone in Children With Skin Grafts After Traumatic Skin Injury: A Randomized Control Trial for Preventative Scar Management
Brief Title: A Randomized Control Trial for Preventative Scar Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-10-134
Record Dates: First submitted 2012-05-10; First posted 2012-05-21 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Hypertrophic Scarring
Keywords: Preventative Scar Management; Skin Grafts; Silicone Therapy; Silicone Pressure Garment Therapy
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silicone Only Therapy (SOT) (Other): Mepiform™ silicone will be utilized by SOT group.
  Interventions: Procedure: Silicone Only Therapy (SOT)
- Silicone Pressure Garment Therapy (SPGT) (Other): Mepiform™ silicone and custom compression garments fabricated by Barton Carey™ will be utilized by SPGT group.
  Interventions: Procedure: Silicone Pressure Garment Therapy (SPGT)

INTERVENTIONS:
Procedure: Silicone Only Therapy (SOT) — SOT group will be instructed to wear the silicone for 23 hours/day, removing only for bathing. A new piece of Mepiform™ silicone should be replaced weekly and applied to clean, dry skin. Compression free medical tape will be used to secure the silicone in place. Patients will be provided with 6 months of topical silicone therapy. If optimal results are achieved prior to 6 months of therapy, the treatment will be discontinued. Patients will also be provided with Scar Management for Skin Grafts Homecare Instructions: Silicone.
  Arms: Silicone Only Therapy (SOT)
Procedure: Silicone Pressure Garment Therapy (SPGT) — SPGT group will be instructed to use the Mepiform™ silicone only for 2 weeks during the interim before final fitting with the custom compression garment. A new piece of Mepiform™ silicone should be replaced weekly and applied to clean, dry skin. The patients will be instructed to wear the silicone for 23 hours/day, removing only for bathing.
  The patient will continue to use the Mepiform™ silicone under the compression garment for the entire length of the study. The garment will be replaced after 3 months of wear, in order to ensure that optimal pressure and silicone management is applied to the area. Patients will be provided with Scar Management for Skin Grafts Homecare Instructions: Silicone and Compression Garment.
  Arms: Silicone Pressure Garment Therapy (SPGT)

SUMMARY:
The study's objective is to compare the global scar outcomes in those treated with silicone only therapy (SOT) versus silicone pressure garment therapy (SPGT) for the prevention of hypertrophic scarring in children with skin grafts after traumatic skin injury.

DETAILED DESCRIPTION:
The goals of this study are to:

1. Examine the difference between patient scores on the POSAS scale in those randomized to silicone pressure garment therapy (SPGT) versus silicone only therapy (SOT) for the prevention of hypertrophic scarring in children with skin grafts after traumatic skin injury at baseline, 8, 16, and 24 weeks.
2. Examine the difference between observer scores on the POSAS scale in those randomized to silicone pressure garment therapy (SPGT) versus silicone only therapy (SOT) for the prevention of hypertrophic scarring in children with skin grafts after traumatic skin injury at baseline, 8, 16, and 24 weeks.
3. Examine the difference between Vancouver scale in those randomized to silicone pressure garment therapy (SPGT) versus silicone only therapy (SOT) for the prevention of hypertrophic scarring in children with skin grafts after traumatic skin injury at baseline, 8, 16, and 24 weeks.
4. Examine the need for surgical intervention in those randomized to silicone pressure garment therapy (SPGT) versus silicone only therapy (SOT) for the prevention of hypertrophic scarring in children with skin grafts after traumatic skin injury.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone surgery within one month prior to enrollment
* patient must have a split-thickness or full thickness skin graft with extremity involvement secondary to a traumatic skin injury (burn, laceration, avulsion or de-gloving type injury) that has healed (based on clinician assessment of wound healing)
* patients with comorbid conditions
* patients must be referred to and attend scar management clinic at DCMC

Exclusion Criteria:

* patients with concave scars at the site of the skin graft
* patients with skin graft scars larger than 4x7 inches
* patients with presence of current skin infection or history of dermatological condition such as eczema
* patients with skin grafts only on parts of the body other than extremities
* patients with reported silicone allergies

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Patient Observer Scar Assessment Scale (POSAS) | Baseline, 8 weeks, 16 weeks, and 24 weeks
  This scale incorporates the patient's/caregiver's perspective on their scar. It measures scar color, pliability, thickness, relief, itching, and pain scored by patient/caregiver. The observer scale measures vascularization, pigmentation, pliability, thickness, and relief.
Vancouver Scar Scale (VSS) | Baseline, 8 weeks, 16 weeks, and 24 weeks
  This scale scores pigmentation, vascularity, pliability, and scar height with the sum of the scores that correlates with hypertrophic scars.

SECONDARY OUTCOMES:
Scar Management Research Intake Form | Baseline through 24 weeks
  This form will include date of enrollment, randomization to group, age, race, gender, date of injury, type of injury, location of injury, type of graft, graft dimensions, date of surgery, date graft healed, number of days for graft to heal, date silicone started, date garment issued, and date silicone/garment discontinued.
Patient Compliance Log (PCL) | Baseline through 24 weeks
  Patients will be given a daily log to record hours of compliance with intervention.
Photographs | Photographs will be collected at each visit (first visit, as well as at weeks 2, 4, 8, 12, 14, 16, 20, and 24
  The Physical/Occupational Therapists are to obtain de-identifiable photographs of the graft site at each visit, in order to have visual documentation of the wound healing process throughout the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Weinfeld, MD, Principal Investigator — Dell Children's Medical Center Rehabilitation Department
Locations (1):
- Dell Children's Medical Center of Central Texas, Austin, Texas, United States